CLINICAL TRIAL: NCT01150565
Title: Phase 1B Pilot Safety Study of LiRIS-TM, A Novel Bladder Drug Delivery Platform in Patients With Interstitial Cystitis
Brief Title: Safety Study of LiRIS in Interstitial Cystitis (IC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: TARIS Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TAR-100-103
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LiRIS low dose (Experimental): The first dose group of approximately 10 patients receive low dose LiRIS on Day 1 to Day 14.
  Interventions: Drug: LiRIS low dose and LiRIS high dose
- LiRIS high dose (Experimental): The second dose group of approximately 10 patients receive high dose LiRIS on Day 1 to Day 14.
  Interventions: Drug: LiRIS low dose and LiRIS high dose

INTERVENTIONS:
Drug: LiRIS low dose and LiRIS high dose — Drug delivery system containing lidocaine; LiRIS (low or high dose) is inserted into bladder via cystoscopy on Day 1 and removed via cystoscopy on Day 14. Designed to release lidocaine over a 14 day period.

SUMMARY:
The purpose of this study is primarily to evaluate the safety and tolerability of two dose levels of an investigational drug-delivery system (LiRIS) in patients who have moderate to severe symptoms of interstitial cystitis.

DETAILED DESCRIPTION:
Approximately 20 female patients with interstitial cystitis will be enrolled in this study at multiple centers in Canada. LiRIS is being developed to provide drug therapy directly into the urinary bladder. LiRIS contains Lidocaine, a marketed drug (approved by Health Canada) which is commonly used for local (skin or oral)anaesthesia. LiRIS is designed to release a controlled amount of lidocaine while in the bladder over a 2 week period.

Two dose groups of approximately 10 patients per group will be enrolled into the study; the first group of patients will receive low dose LiRIS, and the second group will receive high dose LiRIS. All patients receive LiRIS treatment for 14 days, and clinic follow-up at 7 and 14 days after treatment. Additional telephone follow-up occurs at approximately 6 and 10 weeks after LiRIS treatment. The maximum duration of participation, including a screening period of up to 14 days, will be 104 days.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years of age
* If of child-bearing potential, agrees to use effective contraception defined by protocol
* Capable of understanding and completing symptom diaries and questionnaires as required in the study
* Diagnosed with IC, as defined by protocol criteria

Exclusion Criteria:

* Bladder or urethra anatomical feature that, in the opinion of the investigator, might prevent the safe placement, indwelling use, or removal of LiRIS
* History or presence of any medical condition that would interfere with ability to assess symptoms
* Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cystoscopic examination | Days 1 and 14

SECONDARY OUTCOMES:
Bladder pain | During and following treatment; study days 1 to 90

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Nickel, MD, Principal Investigator — Queen's University/Kingston General Hospital
Locations (3):
- Canada (3):
  - Dr. Steinhoff Clinical Research, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax Infirmary, Halifax, Nova Scotia
  - Centre for Applied Urological Research, Kingston, Ontario